CLINICAL TRIAL: NCT02856191
Title: Prospective Study on the Frequency of de Novo Atrial Fibrillation in Septic Shock in Medical Intensive Care
Brief Title: Study on the Frequency of de Novo Atrial Fibrillation in Septic Shock in Medical Intensive Care
Acronym: FACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: QUENOT 2010
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-07

CONDITIONS: Septic Shock; Atrial Fibrillation
MeSH Terms: conditions — Shock, Septic; Atrial Fibrillation

ARMS (1):
- Septic shock (Other)
  Interventions: Other: Holter

INTERVENTIONS:
Other: Holter

SUMMARY:
The aim of this pilot study is to determine, as exhaustively as possible thanks to the continuous and precise recording of heart rhythm, the frequency of de novo atrial fibrillation in septic shock, which is currently unknown, and to identify specific factors that could be associated with the condition. These will be investigated more precisely in a future study. This constitutes the first step in a reflection on the management of Cardiac Arrhythmia by Atrial fibrillation (ACFA) in septic shock in Medical Intensive Care, known as a major prognostic factor for morbimortality, but for which management is uncertain in the absence of reference data.

ELIGIBILITY:
Inclusion Criteria:

* All patients in septic shock (defined as hypotension that is not reversed by fluid resuscitation and requires the use of vasopressor agents) hospitalized in Medical intensive care
* Patients with national health insurance cover
* Age: at least 18 years with no upper limit

Exclusion Criteria:

* Transferred from another intensive care unit for septic shock
* Adults under guardianship
* History of atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation diagnosed on a Holter recording | Over 7 days following the onset of septic shock, or until death or discharge, if one of these events occurs in the 7 days following the onset of the shock.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France